CLINICAL TRIAL: NCT00237627
Title: A Phase I Evaluation of the Combination of Pegylated Liposomal Doxorubicin (Doxil®) With PS-341 in Patients With Refractory Hematologic and Solid Malignancies
Brief Title: Doxorubicin Hydrochloride Liposome and Bortezomib in Treating Patients With Refractory Hematologic Cancer or Malignant Solid Tumor or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 2020; UNC-LCCC-2020; CDR0000368767 (Other: PDQ number)
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Ovarian Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer; recurrent ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia; mast cell leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; atypical chronic myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; chronic myelomonocytic leukemia; refractory hairy cell leukemia; progressive hairy cell leukemia, initial treatment; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; splenic marginal zone lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; primary central nervous system lymphoma; stage III multiple myeloma; stage II multiple myeloma; refractory multiple myeloma; cutaneous B-cell non-Hodgkin lymphoma; recurrent ovarian germ cell tumor; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; unspecified adult solid tumor, protocol specific; recurrent breast cancer; nodal marginal zone B-cell lymphoma
MeSH Terms: conditions — Breast Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Ovarian Neoplasms; Breast Neoplasms, Male; Carcinoma, Ovarian Epithelial; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Mast-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Chronic; Leukemia, Hairy Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Intraocular Lymphoma | interventions — Bortezomib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part 1 (Experimental): Doxil + PS-341
  Interventions: Drug: PS-341; Drug: Doxil
- Part 2 (Experimental): Doxil + Velcade
  Interventions: Drug: Doxil; Drug: Velcade

INTERVENTIONS:
Drug: PS-341 — PS-341 will be administered as an intravenous push into a side arm of either a peripheral or central intravenous line infusing normal saline at 100 ml/hr. Patients will be treated twice weekly for two weeks, followed by a one week rest period, such that the typical days of treatment will be days 1, 4, 8, 11 of each three-week cycle. The initial dose level for PS-341 will be 0.9 mg/m2/dose intravenously, while subsequent dose levels will be determined according to a modified Fibonacci schema
  Arms: Part 1
Drug: Doxil — Doxil will be administered at a dose of 30 mg/m2 as a 1 hour infusion through either a peripheral or central intravenous line every 3 weeks (on day 4 of each 21 day cycle)
  Other Names: pegylated liposomal doxorubicin
Drug: Velcade — Velcade will be adminstered intravenously at 1.3 mg/m2 days 1, 4, 8, 11 every 3 weeks
  Other Names: Bortezomib
  Arms: Part 2

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving doxorubicin hydrochloride liposome together with bortezomib may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of bortezomib when given together with doxorubicin hydrochloride liposome and to see how well they work in treating patients with refractory hematologic cancer or malignant solid tumor or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of bortezomib when administered with pegylated doxorubicin hydrochloride liposome in patients with refractory hematologic or solid tumor malignancies. (Phase I [closed to accrual as of 10/15/2007])
* Determine the dose-limiting toxicity of this regimen in these patients. (Phase I [closed to accrual as of 10/15/2007])
* Determine the response rate in patients with metastatic breast cancer treated with this regimen. (Phase II)

Secondary

* Determine the response in patients with hematologic or solid tumor malignancies treated with this regimen. (Phase I [closed to accrual as of 10/15/2007])
* Determine the time to disease progression in patients with metastatic breast cancer treated with this regimen. (Phase II)
* Obtain further evidence of the safety of this regimen in patients with metastatic breast cancer. (Phase II)

OUTLINE: This is a phase I (closed to accrual as of 10/15/2007), dose-escalation study of bortezomib followed by a phase II study.

* Phase I (closed to accrual as of 10/15/2007): Patients receive bortezomib IV on days 1, 4, 8, and 11 and pegylated doxorubicin hydrochloride liposome IV over 1 hour on day 4. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients receive bortezomib (at the maximum tolerated dose determined in phase I) and pegylated doxorubicin hydrochloride liposome as in phase I.

After completion of study therapy, patients are followed at 1 week.

PROJECTED ACCRUAL: A total of 72 patients will be accrued for the phase I portion of the study and 40 for the phase II portion.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Phase I (closed to accrual as of 10/15/2007)

* Histologically or cytologically confirmed solid tumor or hematologic malignancy, including, but not limited to, any of the following:

  * Breast cancer
  * Ovarian cancer
  * Myeloid or lymphoid leukemia
  * Hodgkin or non-Hodgkin lymphoma
  * Multiple myeloma
* Measurable or evaluable disease
* Must meet 1 of the following criteria:

  * Refractory to at least one prior conventional treatment regimen
  * Not a candidate for conventional therapy
  * No conventional therapy exists
* No clinically or radiographically significant pleural or pericardial effusion

  * Patients with ascites may be eligible at the discretion of the investigator
* Previously treated central nervous system disease allowed provided it has been stable for > 3 months and it is not the only site of measurable disease
* Not eligible for a higher priority protocol

Phase II

* Diagnosis of breast cancer

  * Metastatic disease
* Measurable disease by RECIST criteria
* No symptomatic brain metastases

  * Patients with treated brain metastases that have been stable for > 3 months and does not require chronic steroids are eligible
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Phase I (closed to accrual as of 10/15/2007)

* Karnofsky performance status 60-100%
* Life expectancy ≥ 2 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* WBC ≥ 2,000/mm³
* ANC ≥ 1,500/mm³ (≥ 1,000/mm³ for patients with marrow infiltration)
* Platelet count ≥ 100,000/mm³ (≥ 50,000/mm³ for patients with marrow infiltration)
* Hemoglobin ≥ 8 g/dL
* Creatinine ≤ 2.5 mg/dL OR creatinine clearance ≥ 30 mL/min
* AST and ALT < 2.5 times upper limit of normal (ULN)
* Total bilirubin < 1.2 times ULN
* Prothrombin time (PT) and activated partial thromboplastin time (aPTT) < 1.5 times ULN

  * Patients receiving warfarin or heparin therapy for a history of thrombosis, embolism, or other indication must have PT and/or aPTT within the accepted therapeutic ranges for those indications
* Patients with a history of reactions to other liposomal drug formulations that are not due to the liposome itself may be eligible at the discretion of the investigator
* No known HIV seropositivity
* No known active hepatitis A, B, or C viral infection
* No New York Heart Association class III or IV congestive heart failure
* LVEF ≥ 45% by 2-D ECHO or MUGA
* No acute ischemia or new conduction system abnormality by EKG
* No conduction system abnormality (e.g., left bundle branch block) by EKG that would preclude the ability to detect new ischemic episodes
* No myocardial infarction within the past 6 months
* No significant comorbidity, such as poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that, in the opinion of the investigator, might compromise any aspect of the study
* No uncontrolled infection

  * Patients may have febrile episodes up to 38.5°C if these are felt to be due to tumor fever and the possibility of infection has been ruled out by evaluation
* No prior hypersensitivity reaction to pegylated doxorubicin hydrochloride liposome or doxorubicin hydrochloride

  * Patients with a history of reactions to other liposomal drug formulations and/or to the liposome itself, as opposed to the encapsulated agent, may be excluded at the discretion of the investigator

Phase II

* Female or male
* Menopausal status not specified
* Karnofsky performance status 70-100%
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* Creatinine ≤ 2.5 mg/dL (≤ 200 µmol/L)
* AST and ALT ≤ 2 times ULN
* Alkaline phosphatase ≤ 2 times ULN (unless attributed to tumor)
* Bilirubin ≤ ULN
* Cardiac ejection fraction > 50% by MUGA or 2-D ECHO
* No clinical evidence of congestive heart failure
* No New York Heart Association class II-IV cardiac disease
* No myocardial infarction within the past 6 months
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No evidence of acute ischemia or active conduction system abnormalities by EKG

  * Any EKG abnormality at screening must be documented by the investigator as not medically relevant
* No grade 2 peripheral neuropathy within the past 14 days
* No significant comorbidity that would impair compliance with study therapy or interpretation of study results
* No history of hypersensitivity reactions attributed to a conventional formulation of doxorubicin hydrochloride or the components of pegylated doxorubicin hydrochloride liposome
* No hypersensitivity to bortezomib, boron, or mannitol
* No serious medical or psychiatric illness likely to interfere with participation in this study

PRIOR CONCURRENT THERAPY:

Phase I (closed to accrual as of 10/15/2007)

* More than 3 weeks since prior major surgery
* More than 3 weeks since prior and no concurrent radiotherapy
* More than 4 weeks since prior and no concurrent immunotherapy (i.e., interferon, interleukin, or other cytokine-based treatment)
* More than 3 weeks since prior and no concurrent participation in another therapeutic clinical trial with an experimental drug
* More than 3 weeks since prior and no other concurrent chemotherapy
* No prior doxorubicin dose > 400 mg/m²
* No other concurrent antineoplastic therapy

Phase II

* More than 6 months since prior anthracyclines
* More than 14 days since other prior investigational drugs
* No more than 300 mg/m² of prior doxorubicin or 540 mg/m² of prior epirubicin
* No more than two prior chemotherapy regimens for metastatic disease
* No other concurrent antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2001-05; Primary Completion 2006-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of PS-341 in combination with Doxil (Phase I) | 1 year
  When the current dose level exceeds the MTD, the preceding dose-level will be considered to be the MTD if there have been six patients treated at that dose level. Otherwise, 3 additional patients will be treated at the presumed MTD. No further dose escalation will occur. MTD, like dose limiting toxicity (DLT), will be defined based on toxicities seen within the first cycle. Among the additional 3 patients enrolled in a cohort, if one or more DLT is observed, the MTD will be considered to have been exceeded
Response rate of the combination of Velcade and Doxil in patients with metastatic breast cancer | every 42 days
  Radiographic response will be measured using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Dees, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Robert Z. Orlowski, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Dees EC, O'Neil BH, Lindley CM, Collichio F, Carey LA, Collins J, Riordan WJ, Ivanova A, Esseltine D, Orlowski RZ. A phase I and pharmacologic study of the combination of bortezomib and pegylated liposomal doxorubicin in patients with refractory solid tumors. Cancer Chemother Pharmacol. 2008 Dec;63(1):99-107. doi: 10.1007/s00280-008-0716-8. Epub 2008 Mar 8. PMID 18327587